CLINICAL TRIAL: NCT00748241
Title: An Open Prospective Study to Evaluate the Survival Rate and Marginal Bone Response of Astra Tech Dental Implants, Fixture ST, in Patients With Tooth Loss in the Posterior Maxilla.
Brief Title: Study to Evaluate Implant Survival Rate of Astra Tech Fixture ST in the Posterior Maxilla With One-stage Surgery and Early Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YA-MIC-0002
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-01

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Astra Tech Fixture ST (Experimental)
  Interventions: Device: Astra Tech Fixture ST

INTERVENTIONS:
Device: Astra Tech Fixture ST — Astra Tech Fixture ST Ø 3.5 and 4.5 cm in lengths of 9, 11, 13, 15, 17 and 19 mm.

SUMMARY:
The purpose of this study is primarily to evaluate implant survival rate of Astra Tech Fixture ST placed in the posterior maxilla. A one-stage surgical protocol will be used and the implants will be loaded four weeks after implant installation (early loading). Marginal bone levels, plaque and status of the periimplant mucosa will also be evaluated. The subjects will be followed for three years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75
* Unilateral or bilateral edentulism in the posterior maxilla, last tooth should be the canine or the first bicuspid
* Willing to give informed consent

Exclusion Criteria:

* Bone height < 5 mm, in the planned implant area
* Bone width < 5 mm, in the planned implant area
* Previous bone augmentation procedure in the planned implant area
* Previous failures of endosseous implants
* Untreated caries and/or periodontal disease of residual dentition
* History or presence of any systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* Current alcohol or drug abuse
* Unable or unwilling to return for follow-up visits for 3 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2000-09; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G Valauri, D.D.S., Principal Investigator — New York Dept of Veterans Affairs Medical Center; Michael Toffler, D.D.S., Principal Investigator — New York Dept of Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Dept. of Periodontology, New York Dept of Veterans Affairs Medical Center, New York, New York
  - Dept. of Prosthodontics, New York Dept of Veterans Affairs Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Astra Tech Fixture ST
Started | 19
Completed | 11
Not Completed | 8
Not completed — Implant failure | 1
Not completed — Lost to Follow-up | 5
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Astra Tech Fixture ST
Number analyzed (Participants) | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 61.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival Rate
Description: An implant that has failed to osseointegrate, lost its osseointegration or fractured will be considered a failure effective from the date of removal. Implant Survival Rate will be calculated using the Kaplan-Meier method based on the number of placed implants. Patients who discontinued the study after the last implant failure do not affect the cumulative survival rate.
Time Frame: At follow-up visit: 6 months after implants have been loaded
Population: Population includes subjects who completed the 6 month visit (2 subjects missed the 6 month visit but completed the 1 year visit).
Measure: Number; unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | Astra Tech Fixture ST
Number analyzed (Participants) | 14
Number analyzed (Implants) | 53
Percentage of implants | 89.9

2. Primary Outcome: Implant Survival Rate
Description: An implant that has failed to osseointegrate, lost its osseointegration or fractured will be considered a failure effective from the date of removal. Implant Survival Rate will be calculated using the Kaplan-Meyer method based on the number of placed implants. Patients who discontinued the study after the last implant failure do not affect the cumulative survival rate.
Time Frame: At follow-up visit: 1 year after implants have been loaded
Population: Population includes subjects who completed 12 month visit.
Measure: Number; unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | Astra Tech Fixture ST
Number analyzed (Participants) | 15
Number analyzed (Implants) | 52
Percentage of implants | 89.9

3. Primary Outcome: Implant Survival Rate
Description: as for outcome 2
Time Frame: At follow-up visit: 2 years after implants have been loaded
Population: Population includes subjects who completed 24 month visit.
Measure: Number; unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | Astra Tech Fixture ST
Number analyzed (Participants) | 13
Number analyzed (Implants) | 43
Percentage of implants | 89.9

4. Primary Outcome: Implant Survival Rate
Description: as for outcome 2
Time Frame: At follow-up visit: 3 years after implants have been loaded
Population: Population includes subjects who completed 36 month visit.
Measure: Number; unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | Astra Tech Fixture ST
Number analyzed (Participants) | 11
Number analyzed (Implants) | 39
Percentage of implants | 89.9

5. Secondary Outcome: Implant Failure
Description: Total number of implants reported as failure.
Time Frame: 3 years after implant placement
Population: Number of failed implants based on total number of patients enrolled and total number of placed implants
Measure: Number; unit: Number of implants
Units Other Than Participants: Implants
Arm/Group | Astra Tech Fixture ST
Number analyzed (Participants) | 19
Number analyzed (Implants) | 70
Number of implants | 7

ADVERSE EVENTS:
Arm/Group | Astra Tech Fixture ST
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Astra Tech Fixture ST (N=19)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug overdose (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days